CLINICAL TRIAL: NCT05298488
Title: The Effect of Working at Home Versus at the Office on Risk of Transmission of SARS-CoV-2 and Other Respiratory Agents. A Randomized Controlled Trial
Brief Title: The Effect of Working at Home to Reduce Risk of Respiratory Infection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: The National Institute of Occupational Health, Norway (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CristinID2535463
Record Dates: First submitted 2022-03-07; First posted 2022-03-28 (Actual); Last update posted 2022-03-28 (Actual); Status verified 2022-03

CONDITIONS: Respiratory Tract Infections; COVID-19
Keywords: COVID-19; Infection control; Office from home; Social distancing
MeSH Terms: conditions — Respiratory Tract Infections; COVID-19 | interventions — Working Conditions

STUDY DESIGN:
Intervention Model Description: The participants will be allocated to either office from home for the first four weeks, followed by working at the office for four weeks, or vice versa.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home office for first 4 weeks, and office for the last 4 weeks (Experimental): Participants will work from home for first 4 weeks, and at the office for the last 4 weeks
  Interventions: Behavioral: Home office; Behavioral: Office
- Office for first 4 weeks, and home office for the last 4 weeks (Active Comparator): Participants will work at the office for the first 4 weeks, and from home during the last 4 weeks
  Interventions: Behavioral: Home office; Behavioral: Office

INTERVENTIONS:
Behavioral: Home office — Working from home
Behavioral: Office — Working at the office

SUMMARY:
The researchers will recruit volunteers from various organisations who are willing and able to be randomised to either working from home for 4 weeks followed by working in the office for 4 weeks, or vice versa. The goal is to assess whether working from home has an impact on the risk of symptoms of respiratory infection.

DETAILED DESCRIPTION:
Working in the office entails to various extent contact with colleagues, and for some it includes close contact to others when using public transport to and from work. This likely increases the risk of transmission and many workplaces along with health authorities have strongly advised employees to work from home as much as possible during the COVID-19 pandemic. On the other hand, most people are infected from other family members, and working from home increases exposure to other family members.

There are few, if any trials on the effects of teleworking/home office on the risk of transmission of SARS-CoV-2 and other respiratory agents. Studies that have looked at associations between teleworking and COVID-19 have found a negative correlation.

A systematic review from the National Institute of Occupational Health (STAMI) showed that workers working from home experienced higher work satisfaction and productivity, while also reporting negative effects on work-life balance, professional isolation and working outside core hours. Effects on health outcomes were mixed. The quality of the studies was generally judged as low.

However, working at the office could mean increased exposure to transmission of SARS-CoV-2 and other respiratory agents. Thus, both interventions do pose potential benefits and harms for the participants.

Working from home is a broadly applied intervention nationally and internationally during the COVID-19 pandemic. Establishing what effect this intervention has on actual spread of SARS-CoV-2 and other respiratory agents could hence provide valuable insight to national and local authorities and decision-makers.

The researchers propose to conduct a trial to assess whether working at home impacts on employees' risk of respiratory infection and reduce the risk of work-related outbreaks. The aim is to reject the null hypothesis that working at home does not reduce the risk of respiratory infections or outbreaks among employees.

The researchers plan to conduct the trial as a two-arm multi-period crossover superiority trial where the employees are allocated into two equally sized groups. If this eases the recruitment of firms, the cross-over structure will be dropped.

The first and second arm will cross-over (change treatment) after four weeks. Week 1 and week 5 will be considered run-in periods for these arms, and the data collected these run-in weeks will not be used as outcome data in the statistical analysis.

The plan is to recruit 3-5 large firms with over 2000 eligible participants. Firms located in Oslo and neighbouring municipalities will be included. These are the areas That are seeing the highest incidence rates of SARS-CoV-2 in the ongoing covid-19 pandemic in Norway.

All consenting employees in the selected organizations are eligible to participate in the trial. The organizations can define in advance certain key personnel that cannot take part in the trial.

The investigators will compare the following interventions:

1. Participants will strive to be working from home every day. Participants can go to the office in order to complete tasks that cannot be completed from home.
2. Participants will be working from the office most days, but at least three days a week.

ELIGIBILITY:
Inclusion criteria:

* Over 18 years old
* Employee in a company/organisation that has agreed to let their employees take part
* Willing and able to work form home for 4 weeks (most of the time)

Exclusion crieria:

- Unable to work from home

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Respiratory infection | 8 weeks
  The proportion of participants who report having had symptoms of respiratory disease

SECONDARY OUTCOMES:
COVID-19 | 8 weeks
  Proportion of participants who test positive for SARS-CoV-2 (based on both self-reported and registry data)
Absenteeism | 8 weeks
  Number of days of absence from work.
Secondary cases of respiratory infection | 8 weeks
  Number of secondary cases (transmission from participants in the study) or outbreaks (2 or more cases)
Work-satisfaction | 8 weeks
  Self-reported work-satisfaction (Question: To what extent were you able to carry out your work in a good way during the last week? 5-unit ordinal scale from Very little to Very much).
Work-life balance. | 8 weeks
  Perceived work-life balance (Question: To what extent has your work been at the expense of your own or other family members' free time?) Ordinal 5-unit scale from Very little to Very much.

CONTACTS AND LOCATIONS:
Overall Officials: Atle Fretheim, PhD, Study Director — Head of Centre for Epidemic Interventions Research (CEIR)
Locations (1):
- Norwegian Institute of Public Health, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
The intention is to enable sharing of an anonymised dataset with all interested parties.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: After reporting of the trial findings, estimated to June 2023.